CLINICAL TRIAL: NCT00739973
Title: An 8-week Double-blind, Multicenter, Randomized, Multifactorial, Placebo-controlled, Parallel-group Study to Evaluate the Efficacy and Safety of Aliskiren Administered Alone and in Combination With Amlodipine in Patients With Essential Hypertension
Brief Title: Study to Evaluate the Efficacy and Safety of Aliskiren Alone and in Combination With Amlodipine in Essential Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: CSPA100A2305
Record Dates: First submitted 2008-08-20; First posted 2008-08-22 (Estimated); Results first posted 2011-05-03 (Estimated); Last update posted 2011-06-06 (Estimated); Status verified 2011-06

CONDITIONS: Hypertension
Keywords: Hypertension, Aliskiren, Amlodipine
MeSH Terms: conditions — Hypertension | interventions — aliskiren; Tablets; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (9):
- Placebo (Placebo Comparator): Each dose was to be taken orally with water at approximately 8:00 A.M., except on the morning of the next office/clinic visit, when the study medication was to be taken at the site after the visit procedures were completed. In order to adequately blind the study, patients were required to take a total of 4 tablets and 1 capsule of study medication throughout the study; 5 of the 5 pills taken were placebos.
  Interventions: Drug: Placebo
- Aliskiren 150 mg tablet (Experimental): Each dose was to be taken orally with water at approximately 8:00 A.M., except on the morning of the next office/clinic visit, when the study medication was to be taken at the site after the visit procedures were completed. In order to adequately blind the study, patients were required to take a total of 4 tablets and 1 capsule of study medication throughout the study; 4 of the 5 pills taken were placebos.
  Interventions: Drug: Placebo; Drug: Aliskiren 150 mg tablet
- Aliskiren 300 mg tablet (Experimental): Each dose was to be taken orally with water at approximately 8:00 A.M., except on the morning of the next office/clinic visit, when the study medication was to be taken at the site after the visit procedures were completed. In order to adequately blind the study, patients were required to take a total of 4 tablets and 1 capsule of study medication throughout the study; 4 of the 5 pills taken were placebos.
  Interventions: Drug: Placebo; Drug: Aliskiren 300 mg tablet
- Amlodipine 5 mg capsule (Experimental): Each dose was to be taken orally with water at approximately 8:00 A.M., except on the morning of the next office/clinic visit, when the study medication was to be taken at the site after the visit procedures were completed. In order to adequately blind the study, patients were required to take a total of 4 tablets and 1 capsule of study medication throughout the study; 4 of the 5 pills taken were placebos.
  Interventions: Drug: Placebo; Drug: Amlodipine 5 mg capsule
- Amlodipine 10 mg capsule (Experimental): Each dose was to be taken orally with water at approximately 8:00 A.M., except on the morning of the next office/clinic visit, when the study medication was to be taken at the site after the visit procedures were completed. In order to adequately blind the study, patients were required to take a total of 4 tablets and 1 capsule of study medication throughout the study; 4 of the 5 pills taken were placebos. Amlodipine 10 mg arm starts with 1 week of Amlodipine 5 mg, then force titrated to 10 mg
  Interventions: Drug: Placebo; Drug: Amlodipine 10 mg capsule
- Aliskiren/amlodipine 150/5 mg tablet (Experimental): Each dose was to be taken orally with water at approximately 8:00 A.M., except on the morning of the next office/clinic visit, when the study medication was to be taken at the site after the visit procedures were completed. In order to adequately blind the study, patients were required to take a total of 4 tablets and 1 capsule of study medication throughout the study; 4 of the 5 pills taken were placebos.
  Interventions: Drug: Placebo; Drug: Aliskiren/amlodipine 150/5 mg tablet
- Aliskiren/amlodipine 150/10 mg tablet (Experimental): 150/5 for 1 week, then up-titrated to 150/10 mg. Each dose was to be taken orally with water at approximately 8:00 A.M., except on the morning of the next office/clinic visit, when the study medication was to be taken at the site after the visit procedures were completed. In order to adequately blind the study, patients were required to take a total of 4 tablets and 1 capsule of study medication throughout the study; 4 of the 5 pills taken were placebos.
  Interventions: Drug: Placebo; Drug: Aliskiren/amlodipine 150/10 mg tablet
- Aliskiren/amlodipine 300/5 mg tablet (Experimental): Each dose was to be taken orally with water at approximately 8:00 A.M., except on the morning of the next office/clinic visit, when the study medication was to be taken at the site after the visit procedures were completed. In order to adequately blind the study, patients were required to take a total of 4 tablets and 1 capsule of study medication throughout the study; 4 of the 5 pills taken were placebos.
  Interventions: Drug: Placebo; Drug: Aliskiren/amlodipine 300/5 mg tablet
- Aliskiren/amlodipine 300/10 mg tablet (Experimental): 300/5 for 1 week, then up-titrated to 300/10 mg. Each dose was to be taken orally with water at approximately 8:00 A.M., except on the morning of the next office/clinic visit, when the study medication was to be taken at the site after the visit procedures were completed. In order to adequately blind the study, patients were required to take a total of 4 tablets and 1 capsule of study medication throughout the study; 4 of the 5 pills taken were placebos.
  Interventions: Drug: Placebo; Drug: Aliskiren/amlodipine 300/10 mg tablet

INTERVENTIONS:
Drug: Placebo
Drug: Aliskiren 150 mg tablet
  Arms: Aliskiren 150 mg tablet
Drug: Aliskiren 300 mg tablet
  Arms: Aliskiren 300 mg tablet
Drug: Amlodipine 5 mg capsule
  Arms: Amlodipine 5 mg capsule
Drug: Amlodipine 10 mg capsule
  Arms: Amlodipine 10 mg capsule
Drug: Aliskiren/amlodipine 150/5 mg tablet
  Arms: Aliskiren/amlodipine 150/5 mg tablet
Drug: Aliskiren/amlodipine 150/10 mg tablet
  Arms: Aliskiren/amlodipine 150/10 mg tablet
Drug: Aliskiren/amlodipine 300/5 mg tablet
  Arms: Aliskiren/amlodipine 300/5 mg tablet
Drug: Aliskiren/amlodipine 300/10 mg tablet
  Arms: Aliskiren/amlodipine 300/10 mg tablet

SUMMARY:
Evaluate the efficacy (blood pressure lowering effect) and safety of aliskiren alone and in combination with amlodipine in patients with essential hypertension.

ELIGIBILITY:
Inclusion Criteria:

* msDBP ≥ 90 mmHg and < 110 mmHg at the visit prior to Visit 3 (Visit 2 or optional Visit 201)
* msDBP ≥ 95 mmHg and < 110 mmHg at Visit 3 (Day 1 / randomization).
* All patients must have an absolute difference of ≤ 10 mmHg in their msDBP during the last 2 visits of the single-blind run-in period (Visit 2 and 3 or Visits 201 and 3).

Exclusion Criteria:

* Severe hypertension
* Pregnant or nursing (lactating) women
* Women of child-bearing potential
* Previous or current diagnosis of heart failure (NYHA Class II-IV).
* Serum potassium ≥ 5.3 mEq/L (mmol/L) at Visit 1.
* Uncontrolled Type 1 or Type 2 diabetes mellitus
* Hypersensitivity to renin inhibitors, calcium channel blockers, or to drugs with Similar chemical structures
* History of malignancy within 5 years
* History of hypertensive encephalopathy or cerebrovascular accident, or history of transient ischemic attack (TIA), myocardial infarction, coronary bypass surgery, or any percutaneous coronary intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2694 (Actual)
Dates: Start 2008-09; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Novartis
Locations (18):
- Investigative Site, East Hanover, New Jersey, United States
- Investigative Site, Buenos Aires, Argentina
- Invesigative Site, Canberra, Australia
- Investigative Site, Toronto, Canada
- Investigative Site, Bogotá, Colombia
- Investigative Site, Copenhagen, Denmark
- Investigative Site, Oslo, Finland
- Investigative Site, Athens, Greece
- Investigative Site, Rome, Italy
- Investigative Site, Mexico City, Mexico
- Investigative Site, Panama City, Panama
- Investigative Site, Lima, Peru
- Investigative Site, Bucharest, Romania
- Investigative Site, Moscow, Russia
- Investigative Site, Pretoria, South Africa
- Investigative Site, Madrid, Spain
- Investigative Site, Stockholm, Sweden
- Investigative Site, Taipei, Taiwan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 2694 patients enrolled in the single-blind, placebo run-in period (2 to 4 weeks) of the study. A total of 1688 patients were randomized into the double-blind treatment period (8 weeks). Three patients were mis-randomized, as they were discontinued from the single-blind period and were not treated in the double-blind period.
Groups:
- Placebo: Each dose was to be taken orally with water at approximately 8:00 A.M., except on the morning of the next office/clinic visit, when the study medication was to be taken at the site after the visit procedures were completed. In order to adequately blind the study, patients were required to take a total of 4 tablets and 1 capsule of study medication throughout the study; for this arm all the 5 pills taken were placebos.
- Aliskiren 150 mg; Aliskiren 300 mg; Amlodipine 5 mg; Aliskiren/Amlodipine 150/5 mg; Aliskiren/Amlodipine 300/5 mg: Each dose was to be taken orally with water at approximately 8:00 A.M., except on the morning of the next office/clinic visit, when the study medication was to be taken at the site after the visit procedures were completed. In order to adequately blind the study, patients were required to take a total of 4 tablets and 1 capsule of study medication throughout the study; 4 of the 5 pills taken were placebos.
- Amlodipine 10 mg: Each dose was to be taken orally with water at approximately 8:00 A.M., except on the morning of the next office/clinic visit, when the study medication was to be taken at the site after the visit procedures were completed. In order to adequately blind the study, patients were required to take a total of 4 tablets and 1 capsule of study medication throughout the study; 4 of the 5 pills taken were placebos. Amlodipine 10 mg arm starts with 1 week of Amlodipine 5 mg, then force titrated to 10 mg.
- Aliskiren/Amlodipine 150/10 mg: 150/5 for 1 week, then up-titrated to 150/10 mg. Each dose was to be taken orally with water at approximately 8:00 A.M., except on the morning of the next office/clinic visit, when the study medication was to be taken at the site after the visit procedures were completed. In order to adequately blind the study, patients were required to take a total of 4 tablets and 1 capsule of study medication throughout the study; 4 of the 5 pills taken were placebos.
Period: Single-blind Period (2 to 4 Weeks)
Arm/Group | Placebo | Aliskiren 150 mg | Aliskiren 300 mg | Amlodipine 5 mg | Amlodipine 10 mg | Aliskiren/Amlodipine 150/5 mg | Aliskiren/Amlodipine 150/10 mg | Aliskiren/Amlodipine 300/5 mg | Aliskiren/Amlodipine 300/10 mg Tablet
Started | 2694 (In this period, participants were enrolled to only Placebo arm.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 1685 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1009 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 35 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Abnormal laboratory value(s) | 38 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Abnormal test procedure result(s) | 810 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Patient withdrew consent | 86 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 17 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Administrative problems | 12 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol deviation | 11 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Double-blind:Randomized Period (8 Weeks)
Arm/Group | Placebo | Aliskiren 150 mg | Aliskiren 300 mg | Amlodipine 5 mg | Amlodipine 10 mg | Aliskiren/Amlodipine 150/5 mg | Aliskiren/Amlodipine 150/10 mg | Aliskiren/Amlodipine 300/5 mg | Aliskiren/Amlodipine 300/10 mg Tablet
Started | 198 | 195 (One pt. was mis-randomized, so discontinued from single-blind and was untreated in the double-blind.) | 203 | 185 | 181 | 181 | 183 (2 pts. were mis-randomized, so discontinued from single-blind and were untreated in double-blind.) | 178 | 184
Completed | 168 | 175 | 184 | 173 | 162 | 169 | 170 | 168 | 170
Not Completed | 30 | 20 | 19 | 12 | 19 | 12 | 13 | 10 | 14
Not completed — Adverse Event | 3 | 3 | 1 | 2 | 7 | 3 | 4 | 1 | 4
Not completed — Abnormal laboratory values | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Abnormal test procedure results | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Unsatisfactory therapeutic effect | 17 | 8 | 8 | 4 | 2 | 2 | 1 | 1 | 2
Not completed — Patient no longer needs study drug | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Patient withdrew consent | 4 | 2 | 4 | 3 | 4 | 4 | 3 | 2 | 4
Not completed — Lost to Follow-up | 0 | 2 | 4 | 1 | 2 | 2 | 0 | 3 | 1
Not completed — Administrative problems | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol deviation | 5 | 3 | 1 | 2 | 3 | 1 | 2 | 2 | 3
Not completed — Discont. single-blind, Mis- randomized | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Aliskiren 150 mg | Aliskiren 300 mg | Amlodipine 5 mg | Amlodipine 10 mg | Aliskiren/Amlodipine 150/5 mg | Aliskiren/Amlodipine 150/10 mg | Aliskiren/Amlodipine 300/5 mg | Aliskiren/Amlodipine 300/10 mg Tablet | Total
Number analyzed (Participants) | 198 | 195 | 203 | 185 | 181 | 181 | 183 | 178 | 184 | 1688
Age Continuous [Mean (Standard Deviation); unit: years] | 53.7 (10.32) | 54.3 (11.07) | 54.0 (9.99) | 54.2 (11.61) | 55.0 (10.34) | 53.9 (10.82) | 53.0 (10.59) | 54.8 (10.29) | 54.4 (10.86) | 54.1 (10.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108 | 76 | 108 | 86 | 94 | 84 | 96 | 100 | 78 | 830
  Male | 90 | 119 | 95 | 99 | 87 | 97 | 87 | 78 | 106 | 858

OUTCOME MEASURES:

1. Secondary Outcome: Pairwise Comparison of Aliskiren/Amlodipine 150/5 mg vs. Aliskiren 150 mg on Change in Mean Sitting Systolic Blood Pressure (msSBP)
Description: The arm in which the highest sitting diastolic pressures were found at study entry was the arm used for all subsequent readings. An automated BP measurement device and appropriate size cuff were used to measure arterial sitting blood pressure (BP) at trough with the arm supported at the level of the heart. At each study visit, after having the patient in a sitting position for at least 5 minutes, systolic BP were measured 3 times at 1-2 minute intervals. A mean was calculated from the 3 measurements.
Time Frame: Baseline to end of study (Week 8)
Population: Full Analysis Set (FAS): All participants who were randomized. Participants mis-randomized were excluded from the FAS. Mis-randomized participants refer to participants who were not qualified for randomization but were inadvertently randomized into the study. These participants did not receive study drug.
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Aliskiren 150 mg | Aliskiren/Amlodipine 150/5 mg
Number analyzed (Participants) | 193 | 179
mm Hg | -10.67 (1.01) | -20.64 (1.05)
Statistical Analysis 1: Comparison: Aliskiren 150 mg vs Aliskiren/Amlodipine 150/5 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; A two-way analysis of covariance model with treatment and region as two factors, and the baseline as a covariate; Least Square Mean Difference = -9.97, 95% CI 2-sided [-12.81 to -7.12], Standard Error of Mean 1.45

2. Secondary Outcome: Pairwise Comparison of Aliskiren/Amlodipine 150/5 mg vs. Amlodipine 5 mg on Change in Mean Sitting Systolic Blood Pressure (msSBP)
Description: as for outcome 1
Time Frame: Baseline to end of study (Week 8)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Amlodipine 5 mg | Aliskiren/Amlodipine 150/5 mg
Number analyzed (Participants) | 184 | 179
mm Hg | -15.82 (1.04) | -20.64 (1.05)
Statistical Analysis 1: Comparison: Amlodipine 5 mg vs Aliskiren/Amlodipine 150/5 mg; Test type: Superiority or Other; p = 0.001, ANCOVA; A two-way analysis of covariance model with treatment and region as two factors, and the baseline as a covariate; Least Square mean Difference = -4.82, 95% CI 2-sided [-7.70 to -1.94], Standard Error of Mean 1.47

3. Secondary Outcome: Pairwise Comparison of Aliskiren/Amlodipine 150/5 mg vs. Placebo on Change in Mean Sitting Systolic Blood Pressure (msSBP)
Description: as for outcome 1
Time Frame: Baseline to end of study (Week 8)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Placebo | Aliskiren/Amlodipine 150/5 mg
Number analyzed (Participants) | 198 | 179
mm Hg | -6.79 (1.00) | -20.64 (1.05)
Statistical Analysis 1: Comparison: Placebo vs Aliskiren/Amlodipine 150/5 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; A two-way analysis of covariance model with treatment and region as two factors, and the baseline as a covariate; Least Square Mean Difference = -13.85, 95% CI 2-sided [-16.68 to -11.0], Standard Error of Mean 1.44

4. Secondary Outcome: Pairwise Comparison of Aliskiren/Amlodipine 150/10 mg vs. Aliskiren 150 mg on Change in Mean Sitting Systolic Blood Pressure (mssBP)
Description: as for outcome 1
Time Frame: Baseline to end of study (Week 8)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Aliskiren 150 mg | Aliskiren/Amlodipine 150/10 mg
Number analyzed (Participants) | 193 | 179
mm Hg | -10.67 (1.01) | -23.87 (1.05)
Statistical Analysis 1: Comparison: Aliskiren 150 mg vs Aliskiren/Amlodipine 150/10 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; A two-way analysis of covariance model with treatment and region as two factors, and the baseline as a covariate; Least Square Mean Difference = -13.20, 95% CI 2-sided [-16.04 to -10.4], Standard Error of Mean 1.45

5. Primary Outcome: Pairwise Comparison of Aliskiren/Amlodipine 150/5 mg vs. Aliskiren 150 mg on Change in Mean Sitting Diastolic Blood Pressure (msDBP)
Description: The arm in which the highest sitting diastolic pressures were found at study entry was the arm used for all subsequent readings. An automated BP measurement device and appropriate size cuff were used to measure arterial sitting blood pressure (BP) at trough with the arm supported at the level of the heart. At each study visit, after having the patient in a sitting position for at least 5 minutes, diastolic BP were measured 3 times at 1-2 minute intervals. A mean was calculated from the 3 measurements.
Time Frame: Baseline to end of study (Week 8)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Aliskiren 150 mg | Aliskiren/Amlodipine 150/5 mg
Number analyzed (Participants) | 193 | 179
mm Hg | -7.99 (0.63) | -13.98 (0.66)
Statistical Analysis 1: Comparison: Aliskiren 150 mg vs Aliskiren/Amlodipine 150/5 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; A two-way analysis of covariance model with treatment and region as two factors, and the baseline as a covariate; Least Square Mean Difference = -6.00, 95% CI 2-sided [-7.77 to -4.22], Standard Error of Mean 0.90

6. Primary Outcome: Pairwise Comparison of Aliskiren/Amlodipine 150/5 mg vs. Amlodipine 5 mg on Change in Mean Sitting Diastolic Blood Pressure (msDBP)
Description: as for outcome 5
Time Frame: Baseline to end of study (Week 8)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Amlodipine 5 mg | Aliskiren/Amlodipine 150/5 mg
Number analyzed (Participants) | 184 | 179
mm Hg | -11.0 (0.65) | -13.98 (0.66)
Statistical Analysis 1: Comparison: Amlodipine 5 mg vs Aliskiren/Amlodipine 150/5 mg; Test type: Superiority or Other; p = 0.001, ANCOVA; A two-way analysis of covariance model with treatment and region as two factors, and the baseline as a covariate; Least Square Mean Difference = -2.98, 95% CI 2-sided [-4.77 to -1.19], Standard Error of Mean 0.91

7. Primary Outcome: Pairwise Comparison of Aliskiren/Amlodipine 150/5 mg vs. Placebo on Change in Mean Sitting Diastolic Blood Pressure (msDBP)
Description: as for outcome 5
Time Frame: Baseline to end of study (Week 8)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Placebo | Aliskiren/Amlodipine 150/5 mg
Number analyzed (Participants) | 198 | 179
mm Hg | -5.35 (0.62) | -13.98 (0.66)
Statistical Analysis 1: Comparison: Placebo vs Aliskiren/Amlodipine 150/5 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; A two-way analysis of covariance model with treatment and region as two factors, and the baseline as a covariate; Least Square Mean Difference = -8.63, 95% CI 2-sided [-10.39 to -6.87], Standard Error of Mean 0.90

8. Primary Outcome: Pairwise Comparison of Aliskiren/Amlodipine 150/10 mg vs. Aliskiren 150 mg on Change in Mean Sitting Diastolic Blood Pressure (msDBP)
Description: as for outcome 5
Time Frame: Baseline to end of study (Week 8)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Aliskiren 150 mg | Aliskiren/Amlodipine 150/10 mg
Number analyzed (Participants) | 193 | 179
mm Hg | -7.99 (0.63) | -16.16 (0.66)
Statistical Analysis 1: Comparison: Aliskiren 150 mg vs Aliskiren/Amlodipine 150/10 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; A two-way analysis of covariance model with treatment and region as two factors, and the baseline as a covariate; Least Square Mean Difference = -8.17, 95% CI 2-sided [-9.94 to -6.40], Standard Error of Mean 0.90

9. Primary Outcome: Pairwise Comparison of Aliskiren/Amlodipine 150/10 mg vs. Amlodipine 10 mg on Change in Mean Sitting Diastolic Blood Pressure (msDBP)
Description: as for outcome 5
Time Frame: Baseline to end of study (Week 8)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Amlodipine 10 mg | Aliskiren/Amlodipine 150/10 mg
Number analyzed (Participants) | 179 | 179
mm Hg | -13.82 (0.66) | -16.16 (0.66)
Statistical Analysis 1: Comparison: Amlodipine 10 mg vs Aliskiren/Amlodipine 150/10 mg; Test type: Superiority or Other; p = 0.011, ANCOVA; A two-way analysis of covariance model with treatment and region as two factors, and the baseline as a covariate; Least Sqaure Mean Difference = -2.33, 95% CI 2-sided [-4.14 to -0.53], Standard Error of Mean 0.92

10. Primary Outcome: Pairwise Comparison of Aliskiren/Amlodipine 150/10 mg vs. Placebo on Change in Mean Sitting Diastolic Blood Pressure (msDBP)
Description: as for outcome 5
Time Frame: Baseline to end of study (Week 8)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Placebo | Aliskiren/Amlodipine 150/10 mg
Number analyzed (Participants) | 198 | 179
mm Hg | -5.35 (0.62) | -16.16 (0.66)
Statistical Analysis 1: Comparison: Placebo vs Aliskiren/Amlodipine 150/10 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; A two-way analysis of covariance model with treatment and region as two factors, and the baseline as a covariate; Least Square Mean Difference = -10.81, 95% CI 2-sided [-12.57 to -9.05], Standard Error of Mean 0.90

11. Primary Outcome: Pairwise Comparison of Aliskiren/Amlodipine 300/5 mg vs. Aliskiren 300 mg on Change in Mean Sitting Diastolic Blood Pressure (msDBP)
Description: as for outcome 5
Time Frame: Baseline to end of study (Week 8)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Aliskiren 300 mg | Aliskiren/Amlodipine 300/5 mg
Number analyzed (Participants) | 201 | 175
mm Hg | -10.19 (0.62) | -14.99 (0.66)
Statistical Analysis 1: Comparison: Aliskiren 300 mg vs Aliskiren/Amlodipine 300/5 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; A two-way analysis of covariance model with treatment and region as two factors, and the baseline as a covariate; Least Square Mean Difference = -4.79, 95% CI 2-sided [-6.56 to -3.03], Standard Error of Mean 0.90

12. Primary Outcome: Pairwise Comparison of Aliskiren/Amlodipine 300/5 mg vs. Amlodipine 5 mg on Change in Mean Sitting Diastolic Blood Pressure (msDBP)
Description: as for outcome 5
Time Frame: Baseline to end of study (Week 8)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Amlodipine 5 mg | Aliskiren/Amlodipine 300/5 mg
Number analyzed (Participants) | 184 | 175
mm Hg | -11.0 (0.65) | -14.99 (0.66)
Statistical Analysis 1: Comparison: Amlodipine 5 mg vs Aliskiren/Amlodipine 300/5 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; A two-way analysis of covariance model with treatment and region as two factors, and the baseline as a covariate; Least Square Mean Difference = -3.98, 95% CI 2-sided [-5.78 to -2.18], Standard Error of Mean 0.92

13. Primary Outcome: Pairwise Comparison of Aliskiren/Amlodipine 300/5 mg vs. Placebo on Change in Mean Sitting Diastolic Blood Pressure (msDBP)
Description: as for outcome 5
Time Frame: Baseline to end of study (Week 8)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Placebo | Aliskiren/Amlodipine 300/5 mg
Number analyzed (Participants) | 198 | 175
mm Hg | -5.35 (0.62) | -14.99 (0.66)
Statistical Analysis 1: Comparison: Placebo vs Aliskiren/Amlodipine 300/5 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; A two-way analysis of covariance model with treatment and region as two factors, and the baseline as a covariate; Least Square Mean Difference = -9.64, 95% CI 2-sided [-11.41 to -7.87], Standard Error of Mean 0.90

14. Primary Outcome: Pairwise Comparison of Aliskiren/Amlodipine 300/10 mg vs. Aliskiren 300 mg on Change in Mean Sitting Diastolic Blood Pressure (msDBP)
Description: as for outcome 5
Time Frame: Baseline to end of study (Week 8)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Aliskiren 300 mg | Aliskiren/Amlodipine 300/10 mg Tablet
Number analyzed (Participants) | 201 | 183
mm Hg | -10.19 (0.62) | -16.45 (0.65)
Statistical Analysis 1: Comparison: Aliskiren 300 mg vs Aliskiren/Amlodipine 300/10 mg Tablet; Test type: Superiority or Other; p < 0.001, ANCOVA; A two-way analysis of covariance model with treatment and region as two factors, and the baseline as a covariate; Least Square Mean Difference = -6.26, 95% CI 2-sided [-8.00 to -4.51], Standard Error of Mean 0.89

15. Primary Outcome: Pairwise Comparison of Aliskiren/Amlodipine 300/10 mg vs. Amlodipine 10 mg on Change in Mean Sitting Diastolic Blood Pressure (msDBP)
Description: as for outcome 5
Time Frame: Baseline to end of study (Week 8)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Amlodipine 10 mg | Aliskiren/Amlodipine 300/10 mg Tablet
Number analyzed (Participants) | 179 | 183
mm Hg | -13.82 (0.66) | -16.45 (0.65)
Statistical Analysis 1: Comparison: Amlodipine 10 mg vs Aliskiren/Amlodipine 300/10 mg Tablet; Test type: Superiority or Other; p = 0.004, ANCOVA; A two-way analysis of covariance model with treatment and region as two factors, and the baseline as a covariate; Least Square Mean Difference = -2.63, 95% CI 2-sided [-4.42 to -0.83], Standard Error of Mean 0.92

16. Primary Outcome: Pairwise Comparison of Aliskiren/Amlodipine 300/10 mg vs. Placebo on Change in Mean Sitting Diastolic Blood Pressure (msDBP)
Description: as for outcome 5
Time Frame: Baseline to end of study (Week 8)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Placebo | Aliskiren/Amlodipine 300/10 mg Tablet
Number analyzed (Participants) | 198 | 183
mm Hg | -5.35 (0.62) | -16.45 (0.65)
Statistical Analysis 1: Comparison: Placebo vs Aliskiren/Amlodipine 300/10 mg Tablet; Test type: Superiority or Other; p < 0.001, ANCOVA; A two-way analysis of covariance model with treatment and region as two factors, and the baseline as a covariate; Least Square Mean Difference = -11.10, 95% CI 2-sided [-12.85 to -9.35], Standard Error of Mean 0.89

17. Secondary Outcome: Pairwise Comparison of Aliskiren/Amlodipine 150/10 mg vs. Amlodipine 10 mg on Change in Mean Sitting Systolic Blood Pressure (msSBP)
Description: as for outcome 1
Time Frame: Baseline to end of study (Week 8)
Population: Full Analysis Set (FAS): All randomized patients who received the study medication.
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Amlodipine 10 mg | Aliskiren/Amlodipine 150/10 mg
Number analyzed (Participants) | 179 | 179
mm Hg | -21.04 (1.05) | -23.87 (1.05)
Statistical Analysis 1: Comparison: Amlodipine 10 mg vs Aliskiren/Amlodipine 150/10 mg; Test type: Superiority or Other; p = 0.056, ANCOVA; A two-way analysis of covariance model with treatment and region as two factors, and the baseline as a covariate; Least Square Mean Difference = -2.83, 95% CI 2-sided [-5.73 to -0.07], Standard Error of Mean 1.48

18. Secondary Outcome: Pairwise Comparison of Aliskiren/Amlodipine 150/10 mg vs. Placebo on Change in Mean Sitting Systolic Blood Pressure (msSBP)
Description: as for outcome 1
Time Frame: Baseline to end of study (Week 8)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Placebo | Aliskiren/Amlodipine 150/10 mg
Number analyzed (Participants) | 198 | 179
mm Hg | -6.79 (1.00) | -23.87 (1.05)
Statistical Analysis 1: Comparison: Placebo vs Aliskiren/Amlodipine 150/10 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; A two-way analysis of covariance model with treatment and region as two factors, and the baseline as a covariate; Least Square Mean Difference = -17.08, 95% CI [-19.91 to -14.3], Standard Error of Mean 1.44

19. Secondary Outcome: Pairwise Comparison of Aliskiren/Amlodipine 300/5 mg vs. Aliskiren 300 mg on Change in Mean Sitting Systolic Blood Pressure (msSBP)
Description: as for outcome 1
Time Frame: Baseline to end of study (Week 8)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Aliskiren 300 mg | Aliskiren/Amlodipine 300/5 mg
Number analyzed (Participants) | 201 | 175
mm Hg | -15.37 (0.99) | -21.82 (1.06)
Statistical Analysis 1: Comparison: Aliskiren 300 mg vs Aliskiren/Amlodipine 300/5 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; A two-way analysis of covariance model with treatment and region as two factors, and the baseline as a covariate; Least Square Mean Difference = -6.45, 95% CI 2-sided [-9.29 to -3.62], Standard Error of Mean 1.45

20. Secondary Outcome: Pairwise Comparison of Aliskiren/Amlodipine 300/5 mg vs. Amlodipine 5 mg on Change in Mean Sitting Systolic Blood Pressure (msSBP)
Description: as for outcome 1
Time Frame: Baseline to end of study (Week 8)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Amlodipine 5 mg | Aliskiren/Amlodipine 300/5 mg
Number analyzed (Participants) | 184 | 175
mm Hg | -15.82 (1.04) | -21.82 (1.06)
Statistical Analysis 1: Comparison: Amlodipine 5 mg vs Aliskiren/Amlodipine 300/5 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; A two-way analysis of covariance model with treatment and region asntwo factors, and the baseline as a covariate; Least Square Mean Difference = -6.00, 95% CI 2-sided [-8.90 to -3.11], Standard Error of Mean 1.48

21. Secondary Outcome: Pairwise Comparison of Aliskiren/Amlodipine 300/5 mg vs. Placebo on Change in Mean Sitting Systolic Blood Pressure (msSBP)
Description: as for outcome 1
Time Frame: Baseline to end of study (Week 8)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Placebo | Aliskiren/Amlodipine 300/5 mg
Number analyzed (Participants) | 198 | 175
mm Hg | -6.79 (1.00) | -21.82 (1.06)
Statistical Analysis 1: Comparison: Placebo vs Aliskiren/Amlodipine 300/5 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least Square Mean Difference = -15.03, 95% CI 2-sided [-17.88 to -12.2], Standard Error of Mean 1.45

22. Secondary Outcome: Pairwise Comparison of Aliskiren/Amlodipine 300/10 mg vs. Aliskiren 300 mg on Change in Mean Sitting Systolic Blood Pressure (msSBP)
Description: as for outcome 1
Time Frame: Baseline to end of study (Week 8)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Aliskiren 300 mg | Aliskiren/Amlodipine 300/10 mg Tablet
Number analyzed (Participants) | 201 | 183
mm Hg | -15.37 (0.99) | -23.19 (1.04)
Statistical Analysis 1: Comparison: Aliskiren 300 mg vs Aliskiren/Amlodipine 300/10 mg Tablet; Test type: Superiority or Other; p < 0.001, ANCOVA; A two-way analysis of covariance model with treatment and region as two factors, and the baseline as a covariate; Least Square Mean Difference = -7.82, 95% CI 2-sided [-10.63 to -5.02], Standard Error of Mean 1.43

23. Secondary Outcome: Pairwise Comparison of Aliskiren/Amlodipine 300/10 mg vs. Amlodipine 10 mg on Change in Mean Sitting Systolic Blood Pressure (msSBP)
Description: as for outcome 1
Time Frame: Baseline to end of study (Week 8)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Amlodipine 10 mg | Aliskiren/Amlodipine 300/10 mg Tablet
Number analyzed (Participants) | 179 | 183
mm Hg | -21.04 (1.05) | -23.19 (1.04)
Statistical Analysis 1: Comparison: Amlodipine 10 mg vs Aliskiren/Amlodipine 300/10 mg Tablet; Test type: Superiority or Other; p = 0.143, ANCOVA; A two-way analysis of covariance model with treatment and region as two factors, and the baseline as a covariate; Least Square Mean Difference = -2.16, 95% CI 2-sided [-5.04 to 0.73], Standard Error of Mean 1.47

24. Secondary Outcome: Pairwise Comparison of Aliskiren/Amlodipine 300/10 mg vs. Placebo on Change in Mean Sitting Systolic Blood Pressure (msSBP)
Description: as for outcome 1
Time Frame: Baseline to end of study (Week 8)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Placebo | Aliskiren/Amlodipine 300/10 mg Tablet
Number analyzed (Participants) | 198 | 183
mm Hg | -6.79 (1.00) | -23.19 (1.04)
Statistical Analysis 1: Comparison: Placebo vs Aliskiren/Amlodipine 300/10 mg Tablet; Test type: Superiority or Other; p < 0.001, ANCOVA; A two-way analysis of covariance model with treatment and region as two factors, and the baseline as a covariate; Least Square Mean Difference = -16.40, 95% CI 2-sided [-19.21 to -13.6], Standard Error of Mean 1.43

25. Secondary Outcome: Percentage of Patients With Blood Pressure Control (msSBP < 140 mm Hg and msDBP < 90 mm Hg) at End of Study
Description: Blood pressure control defined as msSBP < 140 mm Hg and msDBP < 90 mm Hg. The arm in which the highest sitting diastolic pressures were found at study entry was the arm used for all subsequent readings. A calibrated sphygmomanometer and appropriate size cuff were used to measure arterial sitting blood pressure (BP) at trough with the arm supported at the level of the heart. At each study visit, after having the patient in a sitting position for at least 5 minutes, systolic/diastolic BP were measured 3 times at 1-2 minute intervals. A mean was calculated from the 3 measurements.
Time Frame: End of study (Week 8)
Population: All patients who were randomized. Following the intent-to-treat principle, patients will be analyzed according to the treatment they were assigned to at randomization. Patients with baseline and Endpoint msDBP values were included in this analysis.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Aliskiren 150 mg | Aliskiren 300 mg | Amlodipine 5 mg | Amlodipine 10 mg | Aliskiren/Amlodipine 150/5 mg | Aliskiren/Amlodipine 150/10 mg | Aliskiren/Amlodipine 300/5 mg | Aliskiren/Amlodipine 300/10 mg Tablet
Number analyzed (Participants) | 198 | 193 | 201 | 184 | 179 | 179 | 179 | 175 | 183
Percentage of Participants | 19.2 | 26.9 | 36.3 | 35.9 | 50.3 | 49.2 | 65.4 | 56.5 | 68.3

26. Secondary Outcome: Percentage of Patients Achieving a Successful Diastolic Blood Pressure Response
Description: Blood pressure response in msDBP is defined as a mean sitting diastolic blood pressure < 90 mmHg or a >=10 mmHg reduction from baseline. A calibrated sphygmomanometer and appropriate size cuff were used to measure arterial sitting blood pressure (BP) at trough with the arm supported at the level of the heart. At each study visit, after having the patient in a sitting position for at least 5 minutes, systolic/diastolic BP were measured 3 times at 1-2 minute intervals. A mean was calculated from the 3 measurements.
Time Frame: End of study (Week 8)
Population: as for outcome 25
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Aliskiren 150 mg | Aliskiren 300 mg | Amlodipine 5 mg | Amlodipine 10 mg | Aliskiren/Amlodipine 150/5 mg | Aliskiren/Amlodipine 150/10 mg | Aliskiren/Amlodipine 300/5 mg | Aliskiren/Amlodipine 300/10 mg Tablet
Number analyzed (Participants) | 198 | 193 | 201 | 184 | 179 | 179 | 179 | 175 | 183
Percentage of Participants | 34.3 | 50.3 | 54.2 | 62.0 | 74.3 | 73.2 | 83.8 | 73.7 | 84.7

27. Secondary Outcome: Percentage of Patients Achieving a Successful Systolic Blood Pressure Response
Description: Blood pressure response in msSBP is defined as a mean sitting systolic blood pressure < 140 mmHg or a >= 20 mmHg reduction from baseline. A calibrated sphygmomanometer and appropriate size cuff were used to measure arterial sitting blood pressure (BP) at trough with the arm supported at the level of the heart. At each study visit, after having the patient in a sitting position for at least 5 minutes, systolic/diastolic BP were measured 3 times at 1-2 minute intervals. A mean was calculated from the 3 measurements.
Time Frame: End of study (Week 8)
Population: as for outcome 25
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Aliskiren 150 mg | Aliskiren 300 mg | Amlodipine 5 mg | Amlodipine 10 mg | Aliskiren/Amlodipine 150/5 mg | Aliskiren/Amlodipine 150/10 mg | Aliskiren/Amlodipine 300/5 mg | Aliskiren/Amlodipine 300/10 mg Tablet
Number analyzed (Participants) | 198 | 193 | 201 | 184 | 179 | 179 | 179 | 175 | 183
Percentage of Participants | 32.3 | 41.5 | 53.2 | 54.9 | 72.1 | 67.6 | 77.1 | 69.7 | 80.3

ADVERSE EVENTS:
Time Frame: Baseline to end of study (Week 8)
Arm/Group | Placebo | Aliskiren 150 mg Tablet | Aliskiren 300 mg Tablet | Amlodipine 5 mg Capsule | Amlodipine 10 mg Capsule | Aliskiren/Amlodipine 150/5 mg Tablet | Aliskiren/Amlodipine 150/10 mg Tablet | Aliskiren/Amlodipine 300/5 mg Tablet | Aliskiren/Amlodipine 300/10 mg Tablet
Serious Adverse Events (participants affected / at risk) | 2/198 | 0/194 | 0/203 | 1/185 | 1/181 | 1/181 | 2/181 | 1/178 | 1/184
Other Adverse Events (participants affected / at risk) | 22/198 | 15/194 | 18/203 | 18/185 | 32/181 | 15/181 | 19/181 | 8/178 | 30/184
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=198) | Aliskiren 150 mg Tablet (N=194) | Aliskiren 300 mg Tablet (N=203) | Amlodipine 5 mg Capsule (N=185) | Amlodipine 10 mg Capsule (N=181) | Aliskiren/Amlodipine 150/5 mg Tablet (N=181) | Aliskiren/Amlodipine 150/10 mg Tablet (N=181) | Aliskiren/Amlodipine 300/5 mg Tablet (N=178) | Aliskiren/Amlodipine 300/10 mg Tablet (N=184)
Retinal detachment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal mass (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=198) | Aliskiren 150 mg Tablet (N=194) | Aliskiren 300 mg Tablet (N=203) | Amlodipine 5 mg Capsule (N=185) | Amlodipine 10 mg Capsule (N=181) | Aliskiren/Amlodipine 150/5 mg Tablet (N=181) | Aliskiren/Amlodipine 150/10 mg Tablet (N=181) | Aliskiren/Amlodipine 300/5 mg Tablet (N=178) | Aliskiren/Amlodipine 300/10 mg Tablet (N=184)
Oedema peripheral (General disorders) | 2 | 2 | 3 | 8 | 25 | 4 | 14 | 2 | 25
Headache (Nervous system disorders) | 20 | 13 | 15 | 11 | 8 | 11 | 8 | 6 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.